CLINICAL TRIAL: NCT02235428
Title: Double-blind, Controlled Trial to Assess the Efficacy of Ipratropium Bromide Associated With High Dose Salbutamol by Repeated Nebulisation Versus Repeat Nebulisation of Salbutamol Alone, for 120 Minutes, in Acute Asthmatic Attacks in Young Children
Brief Title: Study to Assess the Efficacy of Ipratropium Bromide Associated With High Dose Salbutamol by Repeated Nebulisation Versus Repeat Nebulisation of Salbutamol Alone, in Acute Asthmatic Attacks in Young Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 244.2413
Record Dates: First submitted 2014-09-09; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Ipratropium; Albuterol

ARMS (2):
- Ipratropium bromide (Experimental)
  Interventions: Drug: Ipratropium bromide; Drug: Salbutamol
- Salbutamol (Active Comparator)
  Interventions: Drug: Placebo; Drug: Salbutamol

INTERVENTIONS:
Drug: Ipratropium bromide
  Arms: Ipratropium bromide
Drug: Placebo
  Arms: Salbutamol
Drug: Salbutamol

SUMMARY:
To determine whether addition of ipratropium bromide to salbutamol nebulisations produces significantly greater bronchodilation in young children presenting to an emergency department with an acute attack of asthma

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls between 3 and 6 years old
* Presenting to emergency departments with an acute asthmatic attack
* Requiring nebulised bronchodilator therapy
* Rint increased by 200 % compared to theoretical Rint
* Signed, informed consent obtained from the child's parents/legal guardian in accordance with current national legislation and good clinical practice (GCP) defined by the International Conference on Harmonization (ICH)

Exclusion Criteria:

* Ipratropium bromide received within four hours before admission
* First acute asthmatic attack
* Hospital admission to intensive care with asthma within six months before inclusion
* Hospital admission for asthma during the month prior to inclusion
* Corticosteroid-dependent asthma (oral corticosteroid therapy) or recently stopped corticosteroid therapy
* Concomitant cardiac disease
* Life threatening disease requiring immediate management; including: silent chest on auscultation, cyanosis, bradycardia less than 60 beats/min (bpm), confusion, coma
* Hypersensitivity to ipratropium bromide, salbutamol, or to any of their excipients
* Renal or hepatic insufficiency
* Poorly controlled diabetes
* Patients suffering from a disease considered to be severe by the investigator and which, in the opinion of the investigator, could interfere or invalidate the measurements performed in the trial
* Past history of lung surgery
* Major respiratory disease: pulmonary fibrosis, bronchiectasis, sarcoidosis, tuberculosis, respiratory disease due to AIDS, cystic fibrosis
* Patients unable to follow with protocol or correctly undergo the evaluations
* Patients who are taking part in another clinical trial during this trial or who have done so within the month before the trial
* Previous participation in this trial

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 1998-09; Primary Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in pulmonary resistance (Rint) between T0 and T120 | Baseline, 120 minutes after drug administration

SECONDARY OUTCOMES:
Assessment of accessory muscle recruitment on a 4-point scale | Up to 120 minutes after drug administration
Assessment of wheezing on a 4-point scale | Up to 120 minutes after drug administration
Assessment of dyspnoea on a 4-point scale | Up to 120 minutes after drug administration
Changes in respiratory rate | Up to 120 minutes after drug administration
Changes in Oxygen Saturation (ambient air) | Up to 120 minutes after drug administration
Changes in measurement of pulmonary resistance | Up to 120 minutes after drug administration
Number of patients dropped out because of lack of efficacy | Up to 120 minutes after drug administration
Number of patients with adverse events | Up to 17 days after last drug administration
Number of patients dropped out because of adverse events | Up to 17 days after last drug administration
Number of patients with clinical significant findings in blood pressure | Up to 120 minutes after drug administration
Number of patients with clinical significant findings in heart rate | Up to 120 minutes after drug administration
Hospital Admission rate | 120 minutes after drug administration
Assessment of Patient Status by investigator on a 3-question list | 72 hours after drug admimistration